CLINICAL TRIAL: NCT06641713
Title: Hepatic Arterial Infusion Chemotherapy Compared With Transcatheter Arterial Chemoembolizationin Intermediate-advanced Huge Hepatocellular Carcinoma: a Multicenter Retrospective Study
Brief Title: HAIC Compared With TACE in Huge Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Other Study IDs: Liver Projiect 13
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Hepatic Chemotherapy; Liver Cancer
Keywords: Advanced hepatocellular carcinoma; TACE; HAIC; system therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE: TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then conventional TACE or drug-eluting TACE was used.
  Interventions: Procedure: TACE
- HAIC: HIAC was conducted with hepatic arterial infusion of oxaliplatin, fluorouracil, and leucovorin every 3-4 weeks.
  Interventions: Procedure: HAIC

INTERVENTIONS:
Procedure: TACE — TACE was carried out under the guidance of digital subtraction angiography, and hepatic artery angiography was used to assess the location, number, size, and blood supply of the targeted tumor. Then a more selective microcatheter was used to vascularize the tumor. The emulsion of the selected drug and the embolization agents was therefore injected infused into tumor-feeding arteries via the selective microcatheter. A final arteriography confirmed the success of the procedure. The endpoint of the TACE procedure was reached when there was no flow in the tumor-feeding vessels.
  Groups: TACE
Procedure: HAIC — HAIC was carried out under the guidance of digital subtraction angiography, 990and hepatic artery angiography was used to assess the location, number, size, and blood supply of the targeted tumor. Then a more selective microcatheter was used to vascularize the tumor. The FOLFOX regimen was administered via the hepatic artery as follows: 85 or 135 mg/m2 oxaliplatin from hour 0 to 2 on day 1, and 400 mg/m2 leucovorin from hour 2 to 4 on day 1, and 400 mg/m2 fluorouracil bolus at hour 5 on the day 1; and 2400 mg/m2 fluorouracil over 46 h on days 1 and 2. Hepatic arterial infusion chemotherapy administration of oxaliplatin, fluorouracil, and leucovorin via the tumor feeding arteries every 4 weeks
  Groups: HAIC

SUMMARY:
This study intends to compare the efficacy of transcatheter arterial chemical embolization (TACE) with hepatic arterial infusion chemotherapy (HAIC) for patients with intermediate-advanced huge hepatocellular carcinoma.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) and hepatic arterial infusion chemotherapy (HAIC) are effective and safe for hepatocellular carcinoma (HCC). For huge HCC (≥10 cm), the prognosis of this high tumor-burden subtype usually indicates poor outcome and big challenge. TACE is difficult to completely embolize all tumor arteries, so patients have limited benefit from pure hepatic artery embolization. At the same time, excessive embolization will lead to massive tumor necrosis in a short time, and inflammatory necrosis factor will enter the blood, resulting in systemic inflammatory response. HAIC have showed good efficacy especially for advanced huge HCC (≥10 cm) complicated with portal vein tumor thrombus and arteriovenous fistula, and HAIC therapy can be performed with better and higher tumor control.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary HCC.
2. Age between 18 and 75 years;
3. The maximum tumor size ≥10 cm;
4. Intermediate-advanced huge HCC, advanced HCC with PVTT type I-III
5. limited metastases (≤5).
6. Child-Pugh class A or B;
7. Eastern Cooperative Group performance status (ECOG) score of 0-1;
8. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
9. Prothrombin time ≤18s or international normalized ratio < 1.7.

Exclusion Criteria:

1. recurrent HCC;
2. Extrahepatic metastasis >5;
3. Obstructive PVTT involving mesenteric vena cava (PVTT IV).
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
6. Eastern Cooperative Group performance status (ECOG) score of ≥2;
7. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
8. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, observational real-world study to compare the efficacy of HAIC with TACE in advancedhuge hepatocellular carcinoma. This study focused on the management of locoregional therapy . This study will create a database that will provide clinical parameters and outcomes of patients undergoing HIAC and TACE in huge HCC therapy.
Sampling Method: Probability Sample
Enrollment: 664 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months
  ORR, as determined based on tumor response according to mRECIST, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.

SECONDARY OUTCOMES:
Progression-Free-Survival | 12 months
  Progression was defined as progressive disease by independent radiologic review
Overall survival | 24 months
  OS is the length of time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided